CLINICAL TRIAL: NCT01294800
Title: A Phase 2, 12-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Finding Study to Assess the Efficacy and Safety of Preladenant in Japanese Subjects With Moderate to Severe Parkinson's Disease. (Phase 2; Protocol No. P06402)
Brief Title: A Dose Finding Study of Preladenant (SCH 420814) for the Treatment of Parkinson's Disease (PD) in Japanese Patients (P06402)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P06402; MK-3814-026 (Other: Merck)
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Preladenant 2 mg (Experimental): Participants will receive preladenant 2 mg taken orally twice daily (BID), one tablet in the morning and one tablet in the evening, for 12 weeks.
  Interventions: Drug: Preladenant
- Preladenant 5 mg (Experimental): Participants will receive preladenant 5 mg taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
  Interventions: Drug: Preladenant
- Preladenant 10 mg (Experimental): Participants will receive preladenant 10 mg taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
  Interventions: Drug: Preladenant
- Placebo (Placebo Comparator): Participants will receive a placebo to preladenant tablet taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
  Interventions: Drug: Placebo tablet to match Preladenant

INTERVENTIONS:
Drug: Preladenant — 2, 5, or 10 mg tablets taken orally twice daily (BID)
  Other Names: SCH 420814; MK-3814
  Arms: Preladenant 10 mg; Preladenant 2 mg; Preladenant 5 mg
Drug: Placebo tablet to match Preladenant — tablets taken orally BID
  Arms: Placebo

SUMMARY:
This study is to evaluate the efficacy of a range of preladenant doses compared with placebo in participants with moderate to severe Parkinson's disease (PD) experiencing motor fluctuations and receiving a stable dose of levodopa (L-dopa), as measured by "off" time. Participants will continue to receive their stable regimen of L-dopa plus any adjunct medications during the study as prescribed by their physician. Several classes of adjunct medications may be used, including Amantadine, anticholinergics, dopa decarboxylase inhibitors, and dopamine agonists.

Primary Hypothesis: At least the 10 mg twice daily dose of preladenant is superior to placebo as measured by the change from Baseline to Week 12 in the mean "off" time.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of idiopathic PD based on the United Kingdom Parkinson's Disease Society Brain Bank Criteria, judged to be moderate to severe
* Must have received prior therapy with L-dopa for more than 1 year before Screening
* Must have been on a stable, optimal dopaminergic treatment regimen, defined as maximum

therapeutic effect achieved with available anti-Parkinsonian treatment, for at least the 4 weeks immediately before randomization

* If receiving one or more of the following adjunctive treatments: amantadine, anticholinergics, catechol-O-methyltransferase inhibitors, dopa decarboxylase inhibitors, dopamine agonists, entacapone, L-dopa, must have been on a stable regimen of treatment for at least the 4 weeks immediately before randomization
* Hoehn and Yahr stage must be ≥ 2.5 and ≤ 4 following optimum titration of treatment medications at Screening
* Must be experiencing motor fluctuations with or without dyskinesias following optimum titration of

treatment medications and within the 4 weeks immediately before Screening

- Must be experiencing a minimum of 2 hours/day of "off" time as estimated by the investigator

and supported by the symptom diary (Daily Diary) at the Diary Training Visit

- With or without the help of a caregiver, must be capable of maintaining an accurate and

complete symptom diary (Daily Diary) as assessed at the Diary Training Visit

- Must have results of Screening clinical laboratory tests (complete blood count [CBC], blood

chemistries, and urinalysis) within normal limits or clinically acceptable to the investigator at Screening

- Must have results of a physical examination within normal limits or clinically acceptable limits

to the investigator

* Must be able to adhere to dose and visit schedules
* Females of child-bearing potential must have a negative serum pregnancy test (human chorionic

gonadotropin [hCG]) at Screening and must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for 2 weeks after stopping the medication

Exclusion Criteria:

* Must not have a form of drug-induced or atypical parkinsonism, cognitive impairment, bipolar disorder, schizophrenia, or other psychotic disorder
* Must not have had surgery for PD
* Must not have an untreated major depressive disorder meeting Diagnostic and Statistical Manual

of Mental Disorders IV Text Revision (DSM-IV-TR) criteria

- Must not be at imminent risk of self-harm or harm to others, in the investigator's opinion based on

clinical interview

* Must not have participated in any studies using preladenant
* Must not have allergy/sensitivity to preladenant or any of its excipients
* Must not have used any investigational drugs or participated in any other clinical trial within 90 days of Screening

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2011-02-25 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hattori N, Kikuchi M, Adachi N, Hewitt D, Huyck S, Saito T. Adjunctive preladenant: A placebo-controlled, dose-finding study in Japanese patients with Parkinson's disease. Parkinsonism Relat Disord. 2016 Nov;32:73-79. doi: 10.1016/j.parkreldis.2016.08.020. Epub 2016 Aug 27. PMID 27632893

RESULTS

PARTICIPANT FLOW:
Groups:
- Preladenant 2 mg: Participants received preladenant 2 mg taken orally twice daily (BID), one tablet in the morning and one tablet in the evening, for 12 weeks.
- Preladenant 5 mg: Participants received preladenant 5 mg taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
- Preladenant 10 mg: Participants received preladenant 10 mg taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
- Placebo: Participants received a placebo to preladenant tablet taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
Period: Overall Study
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Started | 111 | 113 | 113 | 113
Completed | 100 | 103 | 96 | 97
Not Completed | 11 | 10 | 17 | 16
Not completed — Adverse Event | 7 | 6 | 12 | 5
Not completed — Subject Withdrew Consent | 2 | 2 | 2 | 11
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Non-compliance With Protocol | 0 | 1 | 1 | 0
Not completed — Did Not Meet Protocol Eligibility | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo | Total
Number analyzed (Participants) | 111 | 113 | 113 | 113 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.9) | 67.6 (8.3) | 67.8 (7.6) | 65.8 (9.1) | 67.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 66 | 69 | 64 | 253
  Male | 57 | 47 | 44 | 49 | 197

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean "Off" Time (Hours Per Day) at Week 12
Description: The "on" state is defined as the period of time during which a participant's symptoms of PD improve or disappear following treatment with levodopa (L-dopa) or dopamine agonists. The "off" state is defined as the period of time characterized by the return of symptoms (i..e. tremor, slowness, and rigidity) following treatment with L-dopa or dopamine agonists. Study participants reported their symptoms at half-hour intervals as "off", "on", or "asleep" on their daily diary for 3 days before randomization (baseline) and for the 3 days immediately before their Week-12 visit. The mean change from baseline in "off" time was based on a constrained longitudinal data analysis with treatment, time, and treatment-by-time interaction as fixed effects, and an unstructured covariance matrix was used to model the correlation among repeated measurements.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS) population, which consisted of all randomized participants who received at least one dose of study treatment; had endpoint data subsequent to at least one dose of study treatment; and had baseline data for those analyses requiring baseline data.
Measure: Mean (Standard Deviation); unit: Hours/Day
Groups:
- Preladenant 2 mg: Participants received preladenant 2 mg taken orally BID, one tablet in the morning and one tablet in the evening, for 12 weeks.
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Number analyzed (Participants) | 98 | 101 | 93 | 90
Hours/Day | -1.2 (2.3) | -1.0 (2.6) | -0.9 (2.2) | -0.5 (3.0)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.0564, Constrained longitudinal data analysis; Difference in Least Squares Mean = -0.7, 95% CI 2-sided [-1.37 to 0.02]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.1844, Constrained longitudinal data analysis; Difference in Least Squares Mean = -0.5, 95% CI 2-sided [-1.16 to 0.22]
Statistical Analysis 3: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.3386, Constrained longitudinal data analysis; Difference in Least Squares Mean = -0.3, 95% CI 2-sided [-1.04 to 0.36]

2. Secondary Outcome: Percentage of Participants With ≥30% Reduction in "Off" Time at Week 12
Description: The proportion of responders (≥30% Reduction in "Off" Time at Week 12) was analyzed using a generalized linear mixed model with baseline mean OFF time (hours/day) as a covariate and treatment-by-time interaction as a fixed effect, and an unstructured covariance matrix was used to model the correlation among repeated measurements. Responder rates for each treatment arm are presented as are differences from placebo with 95% confidence interval.
Time Frame: Up to 12 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Number analyzed (Participants) | 110 | 113 | 110 | 112
Percentage of participants | 34.5 | 34.6 | 24.6 | 28.9
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.404, A generalized linear mixed model; Difference in proportions of responders = 5.7, 95% CI 2-sided [-7.75 to 19.00]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.390, A generalized linear mixed model; Difference in proportions of responders = 5.7, 95% CI 2-sided [-7.73 to 18.81]
Statistical Analysis 3: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.508, A generalized linear mixed model; Difference in proportions of responders = -4.9, 95% CI 2-sided [-17.78 to 7.97]

3. Secondary Outcome: Change From Baseline in Mean "On" Time Without Troublesome Dyskinesias (Hours Per Day) at Week 12
Description: When a participant is "on" without dyskinesias, parkinsonian symptoms have dissipated and the participant is experiencing no uncontrollable extraneous movements. Study participants reported their parkinsonian symptoms at half-hour intervals as "off", "on without dyskinesia", "on with non-troublesome dyskinesia", "on with troublesome dyskinesia", or "asleep" on their daily diary for 3 days before randomization and for the 3 days immediately before their Week-12 visit. The mean change from baseline in "on without troublesome dyskinesia" time was based on a constrained longitudinal data analysis with treatment, time, and treatment-by-time interaction as fixed effects, and an unstructured covariance matrix was used to model the correlation among repeated measurements.
Time Frame: Baseline and Week 12
Population: FAS population, which consisted of all randomized participants who received at least one dose of study treatment; had endpoint data subsequent to at least one dose of study treatment; and had baseline data for those analyses requiring baseline data.
Measure: Mean (Standard Deviation); unit: Hours/Day
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Number analyzed (Participants) | 98 | 101 | 93 | 90
Hours/Day | 1.3 (2.5) | 1.0 (2.9) | 1.0 (2.4) | 0.5 (2.9)
Statistical Analysis 1: Comparison: Preladenant 2 mg vs Placebo; Test type: Superiority or Other; p = 0.0509, Constrained longitudinal data analysis; Difference in Least Squares Mean = 0.7, 95% CI 2-sided [-0.00 to 1.43]
Statistical Analysis 2: Comparison: Preladenant 5 mg vs Placebo; Test type: Superiority or Other; p = 0.1847, Constrained longitudinal data analysis; Difference in Least Squares Mean = 0.5, 95% CI 2-sided [-0.23 to 1.19]
Statistical Analysis 3: Comparison: Preladenant 10 mg vs Placebo; Test type: Superiority or Other; p = 0.2021, Constrained longitudinal data analysis; Difference in Least Squares Mean = 0.5, 95% CI 2-sided [-0.25 to 1.19]

4. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to this medicinal product.
Time Frame: Up to 14 weeks
Population: All Participants as Treated population, which included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Number analyzed (Participants) | 111 | 113 | 113 | 113
Participants | 53 | 60 | 69 | 55

5. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to 12 Weeks
Population: All Participants as Treated population, which included all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Number analyzed (Participants) | 111 | 113 | 113 | 113
Participants | 6 | 6 | 12 | 5

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Description: All Participants as Treated population, which included all participants who received at least one dose of study drug
Arm/Group | Preladenant 2 mg | Preladenant 5 mg | Preladenant 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/111 | 5/113 | 7/113 | 3/113
Other Adverse Events (participants affected / at risk) | 19/111 | 23/113 | 25/113 | 14/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=111) | Preladenant 5 mg (N=113) | Preladenant 10 mg (N=113) | Placebo (N=113)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEAT STROKE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
JAW CYST (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
IMPULSE-CONTROL DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACTIVITIES OF DAILY LIVING IMPAIRED (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 2 mg (N=111) | Preladenant 5 mg (N=113) | Preladenant 10 mg (N=113) | Placebo (N=113)
CONSTIPATION (Gastrointestinal disorders) | 3 (3) | 5 (5) | 8 (8) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 5 (5) | 9 (11) | 8 (8) | 8 (10)
FALL (Injury, poisoning and procedural complications) | 8 (10) | 3 (3) | 7 (8) | 0 (0)
DYSKINESIA (Nervous system disorders) | 3 (3) | 7 (7) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication (including, without limitation, slides and texts of oral or other public presentations and texts of any transmission through any electronic media, eg, any computer access system such as the Internet, World Wide Web, etc) that report any results of the trial.